CLINICAL TRIAL: NCT02040155
Title: Real Time In-Vivo Dosimetry For Gynecologic Brachytherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00050297
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Cancer of the Cervix, Cancer of the Endometrium
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Real time dosimetric monitoring of brachytherapy. (Experimental)
  Interventions: Device: Novel nano-scintillator fiber-optic dosimeter (nanoFOD)

INTERVENTIONS:
Device: Novel nano-scintillator fiber-optic dosimeter (nanoFOD) — This is an observational study whose purpose is to determine the feasibility of using a novel nano-scintillator fiber-optic dosimeter (nanoFOD) for the real time dosimetric monitoring of brachytherapy treatment.
  Other Names: nanoFOD

SUMMARY:
This is an observational study. The purpose is to determine the feasibility of using a novel nano-scintillator fiber-optic dosimeter (nanoFOD) for the real time dosimetric monitoring of brachytherapy treatment. Women with gynecologic cancers treated with brachytherapy as part of their standard therapeutic regimen will represent the study population.

DETAILED DESCRIPTION:
Brachytherapy is a curative treatment for many malignancies, brachytherapy delivers a high radiation dose to a very small and well-specified target within a patient with cancer. Yet there is no current convenient, inexpensive, real time method of confirming the radiation dose delivered. There is no current monitoring or fail-safe device for radiation oncologists and their patients if the radiation dose becomes too high, especially to radiation sensitive organs, or conversely if the target receives too little dose.High dose-rate(HDR) brachytherapy is a highly advanced radiation-based cancer treatment, where a very small radioactive source, Iridium-192, is placed in or near the tumor through a catheter or channel. This provides a high radiation dose to the tumor in 5-15 minutes with a precise location, while minimizing radiation exposure to surrounding tissue and organs. This protocol will determine the feasibility of using a novel nano-material based fiber-optic dosimeter (nanoFOD) device, with dimensions less than 1 mm wide, to measure real-time, pin-point, in-vivo radiation dose given during radiation therapy treatments. The size of the device allows placement through a catheter or channel near areas of interest, or within already placed brachytherapy delivery catheters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented neoplasm of the female genital tract.
* Planned brachytherapy as part of standard of care treatment.
* Age > 18 years
* Able to provide and execute informed consent

Exclusion Criteria:

* Any clinical scenario in which the nanoFOD placement or reading would compromise the treatment efficacy, or endanger the patient in any way.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measure dosimetric accuracy of the device with reference to a commercially available dosimeter. | 24 months
  This will only be possible in a subset of women whose implant geometry will result in a radially symmetric dose cloud (i.e. vaginal cylinder cases) so that both the nanoFOD and the reference dosimeter may be placed in a position expected to have the same, or closely similar dose.

SECONDARY OUTCOMES:
Confirm feasibility of clinical application of the nanoFOD for dosimetric monitoring of brachytherapy with complex geometry implants. | 24 months
  Feasibility in this context will mean ease of clinical use (subjective), lack of device failures, and accordance of the nanoFOD dosimetric reading with the planned dose as calculated by the planning software.

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Chino, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States